CLINICAL TRIAL: NCT04499664
Title: Autonomic Cardiovascular Control in Response to Blood Volume Reduction in Blood Donors
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ana-Marija Hristovska, MD, Hvidovre University Hospital
Other Study IDs: H-19069845
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Autonomic Dysfunction; Autonomic Imbalance; Blood Loss
Keywords: Heart rate variabilty; Baroreceptor sensitivity; Autonomic nervous system; Acute blood loss; Blood donors; Autonomic cardiovascular control
MeSH Terms: conditions — Primary Dysautonomias; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 mL of blood stored in a biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood donors: Healhy young male bloddonors, aged 30-45
  Interventions: Device: Monitoring of the autonomic nervous system

INTERVENTIONS:
Device: Monitoring of the autonomic nervous system — Monitoring of the autonomic nervous system using E-patch, LiDCO and Root-Massimo.

SUMMARY:
The function of the autonomic nervous system can be assessed using baroreflex sensitivity (BRS) and heart rate variability (HRV). Decreased HRV has been shown to be predictive of morbidity and mortality in diverse medical conditions such as acute myocardial infarction, aneurysmal subarachnoid haemorrhage, autoimmune diseases, sepsis and surgery.

The function of the autonomic nervous system has not yet been investigated in a "pure hypovolemia" model. The aim of the current study is therefore to investigate and describe the function of the autonomic nervous system prior to, during and after reduction of blood volume in healthy blood donors.

ELIGIBILITY:
Inclusion Criteria:

* Volonteers eligable for blood donation following the Danish legislation
* Male
* Age 30-45
* Written informed consent
* Speak and understand Danish

Exclusion Criteria:

Volonteers not eligable for blood donation following the Danish legislation, among others due to:

* Alcohol and drug abuse
* Cognitive dysfunction
* Use of anxiolytic or antipsychotic drugs
* Arrhythmias or heart failure
* Diabetes mellitus type I
* Diabetes mellitus type II
* Use of opioids
* History of following diseases in the autonomic nervous system: Parkinson disease, multiple sclerosis, autonomic neuropathies
* History of cerebral apoplexy or transitory cerebral ischemia
* Dementia
* American Society of Anesthesiologists (ASA) score ≥ 4

Furthermore:

* History of orthostatic intolerance and/or orthostatic hypotension
* Use of following vasodilator antihypertensive drugs: beta-blockers, angiotensin converting enzyme inhibitors (ACEI), angiotensin 2 receptor blockers (ARBs), calcium channel blockers
* Use of loop diuretics, thiazid diuretics and potassium-sparing diuretics

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male volonteers, aged 30-45, that are eligable for blood donation following the Danish legislation
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in root mean square of successive NN-interval differences (RMSSD) during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in ms

SECONDARY OUTCOMES:
Changes in root mean square of successive NN-interval differences (RMSSD) during sleep | The night before and night after blood donation
  Measured in ms
Changes in standard deviation of N-N intervals (SDNN) during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in ms
Changes in standard deviation of N-N intervals (SDNN) during sleep | The night before and night after blood donation
  Measured in ms
Percentage of successive RR intervals that differ by more than 50 ms (pNN50) during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in %
Percentage of successive RR intervals that differ by more than 50 ms (pNN50) during sleep | The night before and night after blood donation
  Measured in %
Changes in low frequency (LF) power during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in ms^2
Changes in low frequency (LF) power during sleep | The night before and night after blood donation
  Measured in ms^2
Changes high frequency (HF) power during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in ms^2
Changes high frequency (HF) power during sleep | The night before and night after blood donation
  Measured in ms^2
Changes in ratio of LF-to-HF power during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in %
Changes in ratio of LF-to-HF power during sleep | The night before and night after blood donation
  Measured in %
Changes in S (area of the ellipse which represents total HRV) during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in ms
Changes in S (area of the ellipse which represents total HRV) during sleep | The night before and night after blood donation
  Measured in ms
Changes in SD1 (Poincaré plot standard deviation perpendicular the line of identity) during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in ms
Changes in SD1 (Poincaré plot standard deviation perpendicular the line of identity) during sleep | The night before and night after blood donation
  Measured in ms
Changes in SD2 (Poincaré plot standard deviation along the line of identity) during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in ms
Changes in SD2 (Poincaré plot standard deviation along the line of identity) during sleep | The night before and night after blood donation
  Measured in ms
Changes in SD1/SD2 ratio during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in ms
Changes in SD1/SD2 ratio during sleep | The night before and night after blood donation
  Measured in ms
Changes in systolic arterial pressure (SAP) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in mmHg by non-invasive LiDCO
Changes in diastolic arterial pressure (DAP) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in mmHg by non-invasive LiDCO
Changes in mean arterial pressure (MAP) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in mmHg by non-invasive LiDCO
Changes in pulse pressure (PP) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in mmHg by non-invasive LiDCO
Changes in heart rate (HR) during mobilisation | 15 minutes prior to and 15 minutes after blood donation
  Measured in beats min-1 by non-invasive LiDCO
Changes in cardiac output (CO) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in L/min by non-invasive LiDCO
Changes in stroke volume (SV) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in mL by non-invasive LiDCO
Changes in systemic vascular resistance (SVR) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in dynes s cm-5 by non-invasive LiDCO
Changes in cerebral perfusion (ScO2) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in % by Root Masimo
Changes in muscular perfusion (SmO2) during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in % by Root Masimo
Changes in peripheral index during mobilization | 15 minutes prior to and 15 minutes after blood donation
  Measured in % by Root Masimo
Concentration of C-reacitve protein | At time of blood donation
  Measured in gr/dL
V-PLEX Biomarker 54.Plex Kit | Blood taken at time of blood donation
  54 key analytes that are important in inflammation response and immune system regulation as well as numerous other biological processes

OTHER OUTCOMES:
Pain score | 15 minutes prior to and 15 minutes after blood donation
  Measured by verbal rating scale (VRS) 0 - 10 (0 = no pain, 10 = worse pain imaginable) during mobilisation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, Professor, Study Director — Rigshospitalet, Denmark
Locations (1):
- Hvidovre University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Hristovska AM, Uldall-Hansen B, Mehlsen J, Andersen LB, Kehlet H, Foss NB. Orthostatic intolerance after acute mild hypovolemia: incidence, pathophysiologic hemodynamics, and heart-rate variability analysis-a prospective observational cohort study. Can J Anaesth. 2023 Oct;70(10):1587-1599. doi: 10.1007/s12630-023-02556-6. Epub 2023 Sep 26. PMID 37752379